CLINICAL TRIAL: NCT00660738
Title: Comparison of Different Functional Tests and Relation With Functional State and Quality of Life in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Functional Tests in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Bruna Varanda Pessoa, Master Degree, Universidade Federal de Sao Carlos
Other Study IDs: 074/2007
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; walking; exercise test; quality of life; dyspnea; desaturation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 01: Patients with clinical and spirometric diagnosis of COPD, with FEV1<80%

SUMMARY:
Objectives: to evaluate and compare the responses to the various functional tests, and the concordance between the six-minute walk test in hallway (6MWT) and the of oval track (6MWToT), of treadmill (6MWTT), and of treadmill with inclination (6MWTTI), the six-minute step test (6MST) and the sit-to-stand test (STST), in patients with Chronic Obstructive Pulmonary Disease (COPD), and to correlate the responses with functional state and quality of life. Methods: Ten patients with COPD (71±8years, FEV1<80%predicted) were assessed using the functional tests. A dyspnea was assessed using the London Chest Activity of Daily Living and the Medical Research Council scales; and the quality of life was assessed using the St George's Respiratory Questionnaire (SGRQ).

DETAILED DESCRIPTION:
Results: In the interests analysis, there was lower walking distance in the 6MWTT and 6MWTTI was observed, to compare in the 6MWT and 6MWToT; the ΔSp,O2 (delta of arterial oxygen saturation measured by pulse oximeter) in the 6MWTTI was significantly greater that in the 6MWT, but not between to change in dyspnea and fatigue/pain in the lower-limbs between rest and exercise of peak (Δ). Concordance and correlation was observed between the lower Sp,O2 of the 6MWT with the 6MWToT, 6MWTT, 6MWTTI, 6MST and STST. Strong correlations was observed between the performances on the 6MST and 6MWT, 6MWToT and 6MWTT; and between the physical activity domain of the SGRQ with the performances in the 6MWT, 6MWToT, 6MWTT,6MST and STST. Conclusion: The functional tests produced similar subjective responses; however, the 6MWTTI caused greater desaturation that 6MWT. The concordance between the 6MWT and the tests performed, suggests acceptable use of any these tests in the physiotherapeutic clinical routine of the individuals COPD. The tests in performed, except the 6MWTTI, shown to be indicators of the quality of life (physical activity domain).

ELIGIBILITY:
Inclusion Criteria:

* Tiffeneau index<70% e 30%<FEV1<80% predict;
* no presenting exacerbation during the study period;
* clinical stability for the four weeks preceding the study outset;
* no-smokers or ex-smokers.

Exclusion Criteria:

* being incapable of understanding the scales and questionary;
* being unable to perform the tests.

Ages: 55 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic obstructive pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Varanda Pessoa, Master, Physiotherapist, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Special Unit of Respiratory Physiotherapy of Federal University of Sao Carlos (UFSCar), São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Cataneo DC, Kobayasi S, Carvalho LR, Paccanaro RC, Cataneo AJ. Accuracy of six minute walk test, stair test and spirometry using maximal oxygen uptake as gold standard. Acta Cir Bras. 2010 Apr;25(2):194-200. doi: 10.1590/s0102-86502010000200013. PMID 20305888
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] Baarends EM, Schols AM, Mostert R, Wouters EF. Peak exercise response in relation to tissue depletion in patients with chronic obstructive pulmonary disease. Eur Respir J. 1997 Dec;10(12):2807-13. doi: 10.1183/09031936.97.10122807. PMID 9493665
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Cataneo DC, Cataneo AJ. Accuracy of the stair climbing test using maximal oxygen uptake as the gold standard. J Bras Pneumol. 2007 Mar-Apr;33(2):128-33. doi: 10.1590/s1806-37132007000200005. English, Portuguese. PMID 17724530
- [Result] Dal Corso S, Duarte SR, Neder JA, Malaguti C, de Fuccio MB, de Castro Pereira CA, Nery LE. A step test to assess exercise-related oxygen desaturation in interstitial lung disease. Eur Respir J. 2007 Feb;29(2):330-6. doi: 10.1183/09031936.00094006. Epub 2006 Oct 18. PMID 17050559
- [Result] Casanova C, Cote C, Marin JM, Pinto-Plata V, de Torres JP, Aguirre-Jaime A, Vassaux C, Celli BR. Distance and oxygen desaturation during the 6-min walk test as predictors of long-term mortality in patients with COPD. Chest. 2008 Oct;134(4):746-752. doi: 10.1378/chest.08-0520. Epub 2008 Jul 14. PMID 18625667
- [Result] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Result] Casas A, Vilaro J, Rabinovich R, Mayer A, Barbera JA, Rodriguez-Roisin R, Roca J. Encouraged 6-min walking test indicates maximum sustainable exercise in COPD patients. Chest. 2005 Jul;128(1):55-61. doi: 10.1378/chest.128.1.55. PMID 16002916
- [Result] Dourado VZ, Tanni SE, Vale SA, Faganello MM, Sanchez FF, Godoy I. Systemic manifestations in chronic obstructive pulmonary disease. J Bras Pneumol. 2006 Mar-Apr;32(2):161-71. doi: 10.1590/s1806-37132006000200012. English, Portuguese. PMID 17273586
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Hadeli KO, Siegel EM, Sherrill DL, Beck KC, Enright PL. Predictors of oxygen desaturation during submaximal exercise in 8,000 patients. Chest. 2001 Jul;120(1):88-92. doi: 10.1378/chest.120.1.88. PMID 11451821
- [Result] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Result] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Knudson RJ, Lebowitz MD, Holberg CJ, Burrows B. Changes in the normal maximal expiratory flow-volume curve with growth and aging. Am Rev Respir Dis. 1983 Jun;127(6):725-34. doi: 10.1164/arrd.1983.127.6.725. PMID 6859656
- [Result] Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med. 2007 Feb;101(2):286-93. doi: 10.1016/j.rmed.2006.05.007. Epub 2006 Jun 27. PMID 16806873
- [Result] Leung AS, Chan KK, Sykes K, Chan KS. Reliability, validity, and responsiveness of a 2-min walk test to assess exercise capacity of COPD patients. Chest. 2006 Jul;130(1):119-25. doi: 10.1378/chest.130.1.119. PMID 16840391
- [Result] Takigawa N, Tada A, Soda R, Date H, Yamashita M, Endo S, Takahashi S, Kawata N, Shibayama T, Hamada N, Sakaguchi M, Hirano A, Kimura G, Okada C, Takahashi K. Distance and oxygen desaturation in 6-min walk test predict prognosis in COPD patients. Respir Med. 2007 Mar;101(3):561-7. doi: 10.1016/j.rmed.2006.06.017. Epub 2006 Aug 8. PMID 16899358
- [Result] Poulain M, Durand F, Palomba B, Ceugniet F, Desplan J, Varray A, Prefaut C. 6-minute walk testing is more sensitive than maximal incremental cycle testing for detecting oxygen desaturation in patients with COPD. Chest. 2003 May;123(5):1401-7. doi: 10.1378/chest.123.5.1401. PMID 12740254
- [Result] Montes de Oca M, Ortega Balza M, Lezama J, Lopez JM. [Chronic obstructive pulmonary disease: evaluation of exercise tolerance using three different exercise tests]. Arch Bronconeumol. 2001 Feb;37(2):69-74. doi: 10.1016/s0300-2896(01)75017-x. Spanish. PMID 11181240
- [Result] Puente-Maestu L, Garcia de Pedro J, Martinez-Abad Y, Ruiz de Ona JM, Llorente D, Cubillo JM. Dyspnea, ventilatory pattern, and changes in dynamic hyperinflation related to the intensity of constant work rate exercise in COPD. Chest. 2005 Aug;128(2):651-6. doi: 10.1378/chest.128.2.651. PMID 16100150
- [Result] Borel B, Fabre C, Saison S, Bart F, Grosbois JM. An original field evaluation test for chronic obstructive pulmonary disease population: the six-minute stepper test. Clin Rehabil. 2010 Jan;24(1):82-93. doi: 10.1177/0269215509343848. PMID 20053721
- [Result] Oga T, Nishimura K, Tsukino M, Hajiro T, Ikeda A, Mishima M. Relationship between different indices of exercise capacity and clinical measures in patients with chronic obstructive pulmonary disease. Heart Lung. 2002 Sep-Oct;31(5):374-81. doi: 10.1067/mhl.2002.127941. PMID 12487016
- [Result] Brown SE, Casciari RJ, Light RW. Arterial oxygen saturation during meals in patients with severe chronic obstructive pulmonary disease. South Med J. 1983 Feb;76(2):194-8. doi: 10.1097/00007611-198302000-00013. No abstract available. PMID 6823596